CLINICAL TRIAL: NCT04506879
Title: Ultrasound Guided Popliteal Sciatic Nerve Block: Evaluation of Block Dynamics After a Twin Subparaneural Injection Below the Divergence of Common Peroneal and Tibial Nerve.
Brief Title: Popliteal SNB:Evaluation of Block Dynamics After Subparaneural Injection Below CPN & TN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof Manoj K Karmakar, Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CREC.2020.314
Record Dates: First submitted 2020-08-07; First posted 2020-08-10 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Musculoskeletal Diseases or Conditions
Keywords: Popliteal Sciatic nerve block
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Popliteal Sciatic Nerve block (Other): Patients will lie on their chest on the examination couch with both feet rested on the pillow to relax their lower extremity. Ultrasound scan of the nerves in popliteal fossa will be identified and then local anesthetic agents [1.5% lidocaine with 1:200,000 adrenaline and 0.5ml of 8.4% sodium bicarbonate (total 30ml)] will be injected close to the nerves (Common peroneal nerve and tibial nerve). The injections below the bifurcation near the two nerves are expected to produce quicker block than the injections above the bifurcation.
  Interventions: Procedure: Popliteal Sciatic nerve block

INTERVENTIONS:
Procedure: Popliteal Sciatic nerve block — Patients schedule for lower limb surgery under regional anesthesia will receive ultrasound guided subparaneural popliteal sciatic nerve block. After identification of the common peroneal nerve and tibial nerve, local anesthetic agents will be injected close to each nerve below the point of divergence at the popliteal fossa. The spread of the drug and the sensory and motor function of that limb will be assessed regularly till it is ready for surgery.

SUMMARY:
This study aims to assess the effect of twin subparaneural injection into individual paraneural sheaths of Common Peroneal Nerve (CPN) and Tibial Nerve (TN) below their point of divergence from the sciatic nerve on the sensory motor blockade after Popliteal Sciatic Nerve Block (PSNB) at the popliteal fossa (back of the thigh) for patients requiring lower limb surgeries.

DETAILED DESCRIPTION:
Ultrasound (US) guided Popliteal Sciatic Nerve Block (PSNB) has been routinely used to provide surgical anaesthesia for ankle and foot surgeries, and the introduction of ultrasound (US) guidance has improved the ease and accuracy of performing PSNB. However, the challenge of achieving the optimal 'readiness for surgery' time after the US guided PSNB continues to confront anaesthesiologists. Cumulative evidence indicates that a subparaneural PSNB improves sensory motor block outcome when compared to subepimyseal PSNB where the local anaesthetic is deposited outside the paraneural sheath.

While these are encouraging results, producing sensory motor blockade, i.e. surgical anaesthesia in the area innervated by the sciatic nerve within 30 minutes of local anaesthetic (LA) injection, after a subparaneural PSNB, remains a challenge with the success rate varying from 62-92%. Reasons for this shortcoming, despite LA being deposited in subparaneural space, close to the epineurium of the sciatic nerve, is probably multifactorial as the nerve size, surface area exposed to local anaesthetic, and internal architecture (the connective tissue component) of the sciatic nerve and its branches are all seems to influence block onset time and completeness. It was observed from our clinical practice that distal subparaneural injection (twin halo) into individual paraneural sheaths of common peroneal nerve (CPN) and tibial nerve (TN) below the point of divergence at the popliteal fossa demonstrated a faster sensory motor blockade after PSNB. Therefore, this study aims to assess the effect of twin subparaneural injection into individual paraneural sheaths of CPN and TN below their point of divergence from the sciatic nerve on the sensory motor blockade after PSNB at the popliteal fossa.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status I-III scheduled to undergo elective foot and/or ankle surgery under regional anesthesia.

Exclusion Criteria:

* Patient refusal, ASA physical status > Ⅲ, pregnancy, neuromuscular disorder, prior surgery in the popliteal fossa, coagulopathy, allergy to local anaesthetic drugs, and skin infection at the site of needle insertion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-05-27 (Actual); Primary Completion 2023-06-16 (Actual); Study Completion 2023-07-16 (Actual)

PRIMARY OUTCOMES:
the percentage of patients with complete sensory and motor block at 30 min | within 45 minutes after the block (at 5min, 10min, 15min, 20 min, 25min, 30min, 45 min)
  VRS=0 for both sensory and motor score at 30 min. The extent of the sensory blockade will be graded according to VRS (verbal rating scale) for sensory assessment (100 = normal sensation to 0 = no sensation) in the areas innervated by the sciatic nerve. Motor blockade of the deep peroneal nerve (dorsal flexion of the ankle) and tibial nerve (plantar flexion of the ankle) will be graded using a 3-point scale: 2 = normal, 1 = paresis, and 0 = paralysis.

SECONDARY OUTCOMES:
The time taken to complete sensory and motor blockade at 30 min, time to 'readiness for surgery' | within 45 minutes after the block (at 5min, 10min, 15min, 20 min, 25min, 30min, 45min)
  The time point where the sensory block was =< 30 VRS (VRS 0-100, 100=normal sensation and 0= no sensation) and a motor blockade of =< 1 (2=normal, 1=paresis, 0=paralysis),
Success rate of the block | within 45 minutes after the block (at 5min, 10min, 15min, 20min, 25min, 30min, 45min)
  complete abolition of sensation to cold and paralysis of the muscles in the ipsilateral calf and foot
Complication | from immediately after the block till 24 hours afterwards
  any local anesthetic toxicity
Paraesthesia and degree of discomfort | during the block
  Paresthesia (yes or no); degree if discomfort (numeric rating scale 0-100)

CONTACTS AND LOCATIONS:
Overall Officials: Manoj K Karmakar, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Shatin, New Territories, Hong Kong